CLINICAL TRIAL: NCT04268823
Title: A Randomized, Subjects and Investigator Blinded, Placebo Controlled Parallel Group Study to Assess the Mode of Action of QBW251 in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Clinical Study to Assess the Mode of Action of QBW251 in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQBW251B2202
Record Dates: First submitted 2020-01-29; First posted 2020-02-13 (Actual); Results first posted 2023-10-04 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — icenticaftor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- QBW251 (Experimental): Oral use, one capsule twice daily.
  Interventions: Drug: QBW251
- Placebo (Placebo Comparator): Oral use, one capsule twice daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: QBW251 — Capsule 300mg
  Arms: QBW251
Drug: Placebo — Capsule 300mg
  Arms: Placebo

SUMMARY:
The purpose of this study was to determine whether potentiating the cystic fibrosis transmembrane conductance regulator (CFTR) with QBW251 in subjects with COPD would be efficacious with regards to reducing lung and systemic inflammation and bacterial colonization as potential drivers of airway obstruction, airway destruction, remodeling and exacerbations.

Furthermore, this study provided supportive data to investigate the relationship of COPD phenotype and the response in small airway structure, function, mucus load and spirometry indices as well as in improvement of overall COPD symptoms and quality of life.

DETAILED DESCRIPTION:
This was a randomized, subject and investigator blinded, parallel-group, placebo controlled study investigating the mode of action (MoA) and preliminary efficacy and safety of QBW251 administered orally twice daily (b.i.d.) for 12 weeks in subjects with moderate to severe COPD (GOLD 2-3).

The study consisted of the following periods: Screening, Baseline / Day 1, Treatment , and End of the Study followed by an additional post-treatment safety phone call. The total duration for each subject in the study is up to approximately 18 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have signed an Informed Consent Form prior to initiation of any study-related procedure.
2. Male and female adults aged ≥40 years at screening.
3. Patients with stable COPD, stages GOLD 2-3, according to the current GOLD strategy (GOLD 2019) at screening.

   Patients with a post-bronchodilator FEV1/FVC < 0.70 at screening
4. Patients with airflow limitation indicated by a post-bronchodilator FEV1 ≥ 30% and FEV1 < 80% of the predicted normal at Screening who must have had at least 2 documented moderate or at least 1 documented severe exacerbation(s) between January 2019 to study screening.
5. Patients with sputum positive (>0 CFU) for at least one strain of potentially pathogenic microorganism at screening (H influenzae, H parainfluenzae, P aeruginosa, S pneumoniae, S aureus, Moraxella catarrhalis, Enterobacteriaceae, Stenotrophomonas maltophilia, Burkholderia species, and Achromobacter species or any potential pathogenic bacteria measured by dilution/outgrowth. Any organism that is to be included and that is not included in the list of the protocol defined pathogens will be discussed case by case). Sputum samples may be re collected and re-tested once during the screening period.
6. Patients who have been treated with a combination of LABA/LAMA or LABA/ICS or LABA/LAMA/ICS at a stable dose for the last 3 months prior to screening.

   COPD patients are allowed to stay on macrolides as background therapy if they have bronchiectasis as a secondary diagnosis and if they are treated with them at a stable dose 3 months before screening.
7. Patients with plasma fibrinogen level ≥ 320 mg/dL at screening. Fibrinogen may be re-tested once during the screening period.
8. A COPD Assessment Test (CAT) score of at least 10 at screening.
9. Current or ex-smokers who have a smoking history of at least 10 pack years (e.g. 10 pack years = 1 pack/day x 10 years, or 0.5 pack/day x 20 years) at screening.
10. Patients featuring chronic bronchitis, defined as productive cough that occurs on most days (defined as >50% of days) during at least 3 consecutive months in the year prior to screening, as assessed by documentation of patient recollection (anamnesis) or documented in patients' records.
11. Able to communicate well with the investigator, to understand and comply with the requirements of the study.

Exclusion Criteria:

1. Patients with a history of long-QT syndrome or whose QTcF interval at screening (Fridericia method) is prolonged (QTcF >450 ms in males, >460 ms in females).
2. Patients who have a clinically significant* ECG abnormality before randomization. Note: Clinically significant abnormalities may include but are not limited to the following: left bundle branch block, Wolff-Parkinson-White syndrome, clinically significant arrhythmias (e.g., atrial fibrillation, ventricular tachycardia).
3. Clinical laboratory values abnormalities (including Gamma GT, AST, ALT, total bilirubin or creatinine) considered as clinically significant in the opinion of the Investigator at screening. For additional guidance on hepatic parameters see exclusion criterion #5.
4. Patients who have clinically significant renal, cardiovascular (such as but not limited to unstable ischemic heart disease, NYHA Class III/IV left ventricular failure, myocardial infarction), neurological, endocrine, immunological, psychiatric, gastrointestinal, or hematological abnormalities, which could interfere with the assessment of the efficacy and safety of the study treatment, or patients with uncontrolled Type II diabetes.
5. Patients with a history or current treatment for hepatic disease including but not limited to acute hepatitis, cirrhosis or hepatic failure.

   * Patients with stable chronic hepatitis may be included in the study by agreement with Novartis Medical Expert on a case-by-case basis.
   * A history of resolved Hepatitis A is not exclusionary.
   * Patients with prothrombin time international normalized ratio (PT/INR) of more than 1.5xULN at screening. Patients excluded for the PT/INR of more than 1.5xULN can be re-screened when the values have returned to normal.
6. Patients with a history of malignancy of any organ system, treated or untreated, within the past 5 years whether or not there is evidence of local recurrence or metastases, with the exception of localized basal cell carcinoma of the skin. Patients with a history of cancer and 5 years or more disease free survival time may be included in the study by agreement with Novartis Medical Monitor on a case-by-case basis.
7. Patients who develop a COPD exacerbation that required treatment with antibiotics and/or oral corticosteroids and/or hospitalization during screening. Re-screening is permitted after a minimum of 2 weeks after the resolution of the COPD exacerbation (i.e 2 weeks after the stop of SOC therapy for exacerbation).
8. Patients who have had a respiratory tract infection within 4 weeks prior to screening. If a respiratory tract infection occurs during screening, patients can be re-screened after a minimum of 2 weeks after resolution of the respiratory tract infection.
9. Patients with history of asthma or any other clinically relevant lung diseases..
10. Patients with suspected active pulmonary tuberculosis or currently being treatment for active pulmonary tuberculosis.

    Note: Patients with a history of pulmonary tuberculosis can be enrolled if they meet the following requirements: history of appropriate drug treatment followed by negative imaging results within 12 months prior to screening suggesting low probability of recurrent active tuberculosis.
11. Patients with pulmonary lobectomy, lung volume reduction surgery, bronchoscopic lung volume reductions, or lung transplantation.
12. Patients participating in or planning to participate in the active phase of a supervised pulmonary rehabilitation program during the trial. Participation in a maintenance program is permitted. Note: the supervised pulmonary rehabilitation program as a maintenance program has to be ongoing for at least 3 months at the time of enrollment.
13. Patients with a body mass index (BMI) of more than 40 kg/m2.
14. Patients receiving any medications in the classes listed in Table 6-5.
15. Patients receiving any COPD related medications in the classes specified in Table 6-6, unless they undergo the required washout period prior to screening and follow the adjustment to treatment program.
16. Patients receiving medications in the classes listed in Table 6-2 should be excluded unless the medication has been stabilized for the specified period and the stated conditions have been met.
17. Use of other investigational drugs (approved or unapproved) within 30 days or 5 half-lives prior to screening, or until the expected pharmacodynamic effect has returned to baseline (e.g., biologics), whichever is longer; or longer if required by local regulations.
18. Pregnant or nursing (lactating) women, where pregnancy was defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test.
19. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using acceptable effective methods of contraception during study participation.
20. Patients who have not achieved an acceptable spirometry result at screening in accordance with American Thoracic Society (ATS)/ European Respiratory Society (ERS) criteria for acceptability and repeatability.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2022-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (11):
- Novartis Investigative Site, Feldbach, Austria
- Germany (5):
  - Novartis Investigative Site, Heidelberg, Baden-Wurttemberg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Witten
- Switzerland (3):
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Sankt Gallen
  - Novartis Investigative Site, Zurich
- United Kingdom (2):
  - Novartis Investigative Site, Bradford, West Yorkshire
  - Novartis Investigative Site, London

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: Patient Lay Trial Summary — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1578

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 12 investigative sites in 4 countries.
Pre-assignment Details: Informed consent was obtained from each participant in writing at screening before any study specific procedure was performed. The study was explained to the participant by the investigator or designee, who answered any questions, and written information was also provided.
Groups:
- QBW251 300mg: QBW251 300 mg oral dose, one capsule twice daily
- Placebo: Placebo oral dose, one capsule twice daily
Period: Overall Study
Arm/Group | QBW251 300mg | Placebo
Started | 26 | 28
Completed | 24 | 28
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Participant Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | QBW251 300mg | Placebo | Total
Number analyzed (Participants) | 26 | 28 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (7.13) | 67.3 (8.37) | 66.5 (7.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 11 | 27
  Male | 10 | 17 | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 26 | 28 | 54

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Fibrinogen Plasma Concentrations After 12 Weeks of Treatment
Description: To assess the effect of QBW251 compared to placebo after 12 weeks of treatment on fibrinogen. The least-squares means for change from baseline in fibrinogen plasma concentrations after 12 weeks visits for each individual dose group were obtained from a linear mixed effects model for repeated measures (MMRM). A MMRM was fitted to the changes from baseline in fibrinogen for all time points until Day 84. A decrease in fibrinogen plasma concentration indicates improvement.
Time Frame: Baseline, week 12.
Population: Pharmacodynamic (PD) analysis set. Participants were analyzed according to the study treatment received. The PD analysis set included all participants with PD data at both baseline and at least one post-baseline assessment which were not affected by any protocol deviations.
Measure: Least Squares Mean (Standard Error); unit: g/L
Arm/Group | QBW251 300mg | Placebo
Number analyzed (Participants) | 26 | 28
g/L | -0.086 (0.1374) | 0.117 (0.1365)
Statistical Analysis 1: Comparison: QBW251 300mg vs Placebo; Test type: Superiority; p = 0.298, Mixed effects Model for Repeated Measure; Least Squares mean = -0.203, 80% CI 2-sided [-0.524 to 0.119], Standard Error of Mean 0.1938 — Treatment difference (QBW251-placebo)

2. Secondary Outcome: Change From Baseline in Total Bacteria Load of log10 Colony Forming Units (CFU) After 12 Weeks of Treatment
Description: Change from baseline in total bacteria load of colony forming units of potentially pathogenic microorganisms in sputum. A decrease in airway bacterial colonization as detected in the sputum is considered improvement.
Time Frame: Baseline, week 12.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: log10 CFU/mL
Arm/Group | QBW251 300mg | Placebo
Number analyzed (Participants) | 26 | 28
log10 CFU/mL | -0.2 (0.30) | 0.0 (0.32)
Statistical Analysis 1: Comparison: QBW251 300mg vs Placebo; Test type: Superiority; p = 0.651, Mixed effects Model for Repeated Measure; Least Squares mean = -0.2, 80% CI 2-sided [-0.9 to 0.5], Standard Error of Mean 0.44 — Treatment difference (QBW251-placebo)

3. Secondary Outcome: Change From Baseline in COPD Assessment Test (CAT) Questionnaire After 12 Weeks of Treatment
Description: The COPD assessment test (CAT) is a short instrument which was used to quantify the symptom burden of COPD and disease severity of participants in this study. The CAT consists of 8 items, each presented as a semantic 6-point differential scale (0-5), providing a total range from 0 to 40. A higher score indicates a worse health status.
Time Frame: Baseline, week 12.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | QBW251 300mg | Placebo
Number analyzed (Participants) | 26 | 28
Score on a scale | -3.55 (0.947) | -2.16 (0.874)
Statistical Analysis 1: Comparison: QBW251 300mg vs Placebo; Test type: Superiority; p = 0.288, Mixed effects Model for Repeated Measure; Least Squares mean = -1.39, 80% CI 2-sided [-3.55 to 0.78], Standard Error of Mean 1.290 — Treatment difference (QBW251-placebo)

4. Secondary Outcome: Change From Baseline in Euro Quality of Life-5 Dimensions-3 Level (EQ-5D-3L) Questionnaire After 12 Weeks of Treatment
Description: The EQ-5D-3L questionnaire is a general health status and health utility measure which captures 5 dimensions of health state: mobility, self-care, usual activities, pain/discomfort and anxiety/depression and visual analog has a scale 0 to 100 (0=worst imaginable health state, 100=best imaginable health state).
Time Frame: Baseline, week 12.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | QBW251 300mg | Placebo
Number analyzed (Participants) | 26 | 28
Score on a scale | 7.63 (3.116) | 3.43 (2.854)
Statistical Analysis 1: Comparison: QBW251 300mg vs Placebo; Test type: Superiority; p = 0.338, Mixed effects Model for Repeated Measure; Least Squares mean = 4.20, 80% CI 2-sided [-3.09 to 11.48], Standard Error of Mean 4.336 — Treatment difference (QBW251-placebo)

5. Secondary Outcome: Change From Baseline in St. George's Respiratory Questionnaire (SGRQ) Total and Domain Scores After 12 Weeks of Treatment
Description: The St. George's Respiratory questionnaire (SGRQ) was used to provide the health status measurements. The SGRQ contains 50 items divided into two parts covering three aspects of health related to COPD: Part I covers "Symptoms", Part II covers "Activity" and "Impacts". A score is calculated for each of these three subscales including the "Total" score. In each case the lowest possible value is zero and the highest 100. Higher values correspond to greater impairment of health status.
Time Frame: Baseline, week 12.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | QBW251 300mg | Placebo
Number analyzed (Participants) | 26 | 28
Score on a scale
  Week 12- total score | -2.99 (2.297) | -2.17 (2.111)
  Week 12- Symptoms score | -0.98 (3.052) | -6.73 (2.806)
  Week 12- Activity score | -1.96 (2.388) | -1.35 (2.194)
  Week 12- Impact score | -3.72 (2.944) | -1.65 (2.705)
Statistical Analysis 1: Comparison: QBW251 300mg vs Placebo; Total score; Test type: Superiority; p = 0.795, Mixed effects Model for Repeated Measure; Least Squares mean = -0.82, 80% CI 2-sided [-6.05 to 4.42], Standard Error of Mean 3.147 — Treatment difference (QBW251-placebo)
Statistical Analysis 2: Comparison: QBW251 300mg vs Placebo; Symptoms score; Test type: Superiority; p = 0.170, Mixed effects Model for Repeated Measure; Least Squares mean = 5.75, 80% CI 2-sided [-1.16 to 12.66], Standard Error of Mean 4.155 — Treatment difference (QBW251-placebo)
Statistical Analysis 3: Comparison: QBW251 300mg vs Placebo; Activity score; Test type: Superiority; p = 0.851, Mixed effects Model for Repeated Measure; Least Squares mean = -0.61, 80% CI 2-sided [-6.02 to 4.80], Standard Error of Mean 3.259 — Treatment difference (QBW251-placebo)
Statistical Analysis 4: Comparison: QBW251 300mg vs Placebo; Impact score; Test type: Superiority; p = 0.610, Mixed effects Model for Repeated Measure; Least Squares mean = -2.07, 80% CI 2-sided [-8.78 to 4.65], Standard Error of Mean 4.035 — Treatment difference (QBW251-placebo)

6. Secondary Outcome: Change From Baseline in Cough and Sputum Assessment Questionnaire (CASA-Q) After 12 Weeks of Treatment
Description: The CASA-Q is a validated questionnaire used to measure cough and sputum production, and their impact in patients with COPD and/or chronic bronchitis. There are only domain scores and no overall score. The scores in each domain range from 0 to 100, with lower scores indicating more severe symptoms or a higher impact.
Time Frame: Baseline, week 12.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | QBW251 300mg | Placebo
Number analyzed (Participants) | 26 | 28
Score on a scale
  Week 12 - cough symptom score | 4.36 (3.339) | 4.11 (3.083)
  Week 12 - sputum symptom score | 5.00 (3.401) | 0.78 (3.121)
  Week 12 - cough impact score | 4.64 (2.936) | 2.60 (2.697)
  Week 12 - sputum impact score | 3.22 (3.298) | 2.28 (3.017)
Statistical Analysis 1: Comparison: QBW251 300mg vs Placebo; Cough symptom score; Test type: Superiority; p = 0.956, Mixed effects Model for Repeated Measure; Least Squares mean = 0.25, 80% CI 2-sided [-7.30 to 7.80], Standard Error of Mean 4.557 — Treatment difference (QBW251-placebo)
Statistical Analysis 2: Comparison: QBW251 300mg vs Placebo; Sputum symptom score; Test type: Superiority; p = 0.369, Mixed effects Model for Repeated Measure; Least Squares mean = 4.22, 80% CI 2-sided [-3.55 to 11.99], Standard Error of Mean 4.671 — Treatment difference (QBW251-placebo)
Statistical Analysis 3: Comparison: QBW251 300mg vs Placebo; Cough impact score; Test type: Superiority; p = 0.613, Mixed effects Model for Repeated Measure; Least Squares mean = 2.03, 80% CI 2-sided [-4.61 to 8.68], Standard Error of Mean 4.001 — Treatment difference (QBW251-placebo)
Statistical Analysis 4: Comparison: QBW251 300mg vs Placebo; Sputum impact score; Test type: Superiority; p = 0.835, Mixed effects Model for Repeated Measure; Least Squares mean = 0.94, 80% CI 2-sided [-6.58 to 8.47], Standard Error of Mean 4.518 — Treatment difference (QBW251-placebo)

7. Secondary Outcome: Pre-dose Trough Concentration (Ctrough) of QBW251
Description: Pharmacokinetic blood samples were collected and evaluated in all participants exposed to QBW251. QBW251 was analyzed by a validated Liquid Chromatography with tandem Mass Spectrometry. Concentration below the lower limit of quantification (LLOQ) was reported as zero.
Time Frame: Day 1, Day 28, Day 56 and Day 84
Population: The PK analysis set included all participants with at least one available valid (i.e., not flagged for exclusion) PK concentration measurement, who received QBW251 and experienced no protocol deviations with relevant impact on PK data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | QBW251 300mg
Number analyzed (Participants) | 26
ng/mL
  Day 1: number analyzed (Participants) | 23
  Day 1 | 0.00 (0.00)
  Day 28: number analyzed (Participants) | 22
  Day 28 | 526 (735)
  Day 56: number analyzed (Participants) | 23
  Day 56 | 489 (540)
  Day 84: number analyzed (Participants) | 24
  Day 84 | 567 (883)

8. Secondary Outcome: Change From Baseline in Trough FEV1 After 12 Weeks of Treatment
Description: FEV1 (forced expiratory volume in one second) is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation, measured through spirometry testing. The least-squares means for change from baseline in FEV1 to assess the effect of QBW251 compared to placebo after 12 weeks were obtained from a linear mixed effects model for repeated measures (MMRM). A positive change from baseline in pre-dose FEV1 is considered a favourable outcome.
Time Frame: Baseline, week 12.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: liters (L)
Arm/Group | QBW251 300mg | Placebo
Number analyzed (Participants) | 26 | 28
liters (L) | 0.0 (0.03) | -0.1 (0.03)
Statistical Analysis 1: Comparison: QBW251 300mg vs Placebo; Test type: Superiority; p = 0.335, Mixed effects Model for Repeated Measure; Least Squares Mean = 0.0, 80% CI 2-sided [0.0 to 0.1], Standard Error of Mean 0.04 — Treatment difference (QBW251-placebo)

9. Secondary Outcome: Change From Baseline in FVC After 12 Weeks of Treatment
Description: To assess the effect of QBW251 compared to placebo after 12 weeks of treatment on spirometry (Forced Vital Capacity). Forced Vital Capacity (FVC) is the amount of air which can be forcibly exhaled from the lungs after taking the deepest breath possible.
Time Frame: Baseline, week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: liters (L)
Arm/Group | QBW251 300mg | Placebo
Number analyzed (Participants) | 26 | 28
liters (L) | -0.1 (0.05) | -0.1 (0.05)
Statistical Analysis 1: Comparison: QBW251 300mg vs Placebo; Test type: Superiority; p = 0.645, Mixed effects Model for Repeated Measure; Least Squares mean = 0.0, 80% CI 2-sided [-0.1 to 0.1], Standard Error of Mean 0.07 — Treatment difference (QBW251-placebo)

10. Secondary Outcome: Change From Baseline in FEV1/FVC After 12 Weeks of Treatment
Description: To assess the effect of QBW251 compared to placebo after 12 weeks of treatment on spirometry. FEV1/FVC is the percent of a person's vital capacity that they are able to expire in the first second of forced expiration (FEV1) to the full, forced vital capacity (FVC).
Time Frame: Baseline, week 12.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | QBW251 300mg | Placebo
Number analyzed (Participants) | 26 | 28
percent | 1.7 (0.58) | -0.3 (0.55)
Statistical Analysis 1: Comparison: QBW251 300mg vs Placebo; Test type: Superiority; p = 0.010, Mixed effects Model for Repeated Measure; Least Squares mean = 2.1, 80% CI 2-sided [0.8 to 3.4], Standard Error of Mean 0.80 — Treatment difference (QBW251-placebo)

11. Secondary Outcome: Maximum Observed Plasma Concentrations (Cmax) of QBW251 in a Subset of Patient Population
Description: Cmax is the maximum (peak) observed plasma concentration of QBW251 after dose administration. QBW251 was analyzed by a validated Liquid Chromatography with tandem Mass Spectrometry. Concentration below the lower limit of quantification was reported as zero.
  Serial plasma PK concentrations were sampled on Day 1 and Day 28 up to 8 hours post dose in a subset of the patient population.
Time Frame: Pre dose, Post dose (1, 2, 3, 4, 6, and 8 hours) at Day 1 and Day 28.
Population: The PK analysis set included all participants with at least one available valid (i.e., not flagged for exclusion) PK concentration measurement, who received QBW251 and experienced no protocol deviations with relevant impact on PK data. The analysis was performed on a subset of the PK analysis set for participants where serial plasma PK concentrations were sampled.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | QBW251 300mg
Number analyzed (Participants) | 12
ng/mL
  Day 1 | 1000 (608)
  Day 28 | 1580 (866)

12. Secondary Outcome: Maximum Observed Plasma Concentrations (Cmax) of QBW251
Description: Cmax is the maximum (peak) observed plasma concentration of QBW251 after dose administration. QBW251 was analyzed by a validated Liquid Chromatography with tandem Mass Spectrometry. Concentration below the lower limit of quantification was reported as zero.
  On Day 56 and Day 84 pre-dose and 3 hour post dose sparse samples were collected from all participants.
Time Frame: Post-dose (3 hours) at Day 56 and Day 84.
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | QBW251 300mg
Number analyzed (Participants) | 21
ng/mL
  Day 56: number analyzed (Participants) | 20
  Day 56 | 903 (648)
  Day 84 | 997 (497)

13. Secondary Outcome: Area Under Plasma Concentration-time Curve From Time Zero to the Last Measurable Concentration Sampling Time (AUClast) of QBW251
Description: Pharmacokinetic blood samples were collected and evaluated in all participants exposed to QBW251. QBW251 was analyzed by a validated Liquid Chromatography with tandem Mass Spectrometry. Concentration below the lower limit of quantification was reported as zero. AUClast is the area under the plasma concentration-time curve from time zero to the time of last quantifiable concentration (tlast) of QBW251.
Time Frame: Pre dose, Post dose (1, 2, 3, 4, 6, and 8 hours) at Day 1 and Day 28
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | QBW251 300mg
Number analyzed (Participants) | 12
h*ng/mL
  Day 1 | 4290 (3630)
  Day 28 | 7320 (5950)

14. Secondary Outcome: On-treatment Analysis of Time to First COPD Exacerbation Using Cox Regression Model
Description: To assess the effect of QBW251 compared to placebo after 12 weeks of treatment on COPD exacerbations, exacerbations defined by EXACT-PRO questionnaire. The protocol defined that the time-to-event analyses were to be carried out only upon sufficient number of exacerbation events occur during the study to estimate the median in either of the treatment groups.
Time Frame: Baseline, week 12.
Population: No patients analyzed as there was not a sufficient number of exacerbations to carry out the time to event analysis.
Arm/Group | QBW251 300mg | Placebo
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Proportion of Patients (Percentage) With Exacerbations
Description: The EXACT-PRO is a validated 14-item electronic questionnaire designed to detect the frequency, severity, and duration of exacerbations in participants with COPD. Minimum score is 0 and Maximum score is 40 (higher scores indicate worsening indicative of an exacerbation). EXACT-PRO-defined exacerbations are defined as a persistent increase from baseline in total EXACT-PRO score of ≥9 points for 3 days or ≥12 points for 2 days.
Time Frame: From first dose of study treatment until last dose of study treatment plus 7 days, up to a maximum duration of 99 days
Population: Due to study termination with fewer enrollment of subjects, and shorter treatment duration (i.e., 12 weeks), statistical summaries were not performed as unlikely to provide meaningful values.
Measure: Count of Participants; unit: Participants
Arm/Group | QBW251 300mg | Placebo
Number analyzed (Participants) | 26 | 28
Participants | 3 | 3

16. Secondary Outcome: Annualized Rate of EXACT-PRO-defined Exacerbations
Description: The Exacerbations of COPD Tool-Patient Reported Outcome (EXACT-PRO) is a validated 14-item electronic questionnaire designed to detect the frequency, severity, and duration of exacerbations in participants with COPD. Minimum score is 0 and Maximum score is 40 (higher scores indicate worsening indicative of an exacerbation). EXACT-PRO-defined exacerbations are defined as a persistent increase from baseline in total EXACT-PRO score of ≥9 points for 3 days or ≥12 points for 2 days. Annualized rate of exacerbations was analyzed using a generalized linear model assuming a negative binomial distribution.
Time Frame: From first dose of study treatment until last dose of study treatment plus 7 days, up to a maximum duration of 99 days
Population: as for outcome 1
Measure: Number (80% Confidence Interval); unit: exacerbations per participant per year
Arm/Group | QBW251 300mg | Placebo
Number analyzed (Participants) | 24 | 28
exacerbations per participant per year | 1.22 [0.74 to 2.03] | 1.01 [0.61 to 1.67]

17. Secondary Outcome: Change From Baseline in Airway Wall and Lumen
Description: To assess the effect of QBW251 compared to placebo after 12 weeks of treatment on airway structure and function, measured by High Resolution Computed Tomography (HRCT).
Time Frame: Baseline, week 12.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | QBW251 300mg | Placebo
Number analyzed (Participants) | 21 | 18
mm
  Lung, Left, Inferior Lobe, Posterior Basal Segment | 0.01 (0.201) | 0.02 (0.155)
  Lung, Left, Superior Lobe, Apical Segment | -0.01 (0.150) | 0.06 (0.134)
  Lung, Right, Inferior Lobe, Posterior Basal Segment: number analyzed (Participants) | 19 | 18
  Lung, Right, Inferior Lobe, Posterior Basal Segment | 0.08 (0.378) | -0.03 (0.149)
  Lung, Right, Middle Lobe, Lateral Segment: number analyzed (Participants) | 20 | 17
  Lung, Right, Middle Lobe, Lateral Segment | 0.00 (0.145) | -0.06 (0.105)
  Lung, Right, Superior Lobe, Apical Segment | -0.02 (0.128) | 0.02 (0.092)

18. Secondary Outcome: Change From Baseline in Percent Global and Regional Air Trapping After 12 Weeks of Treatment
Description: To assess the effect of QBW251 compared to placebo after 12 weeks of treatment on airway structure and functions, measured by High Resolution Computed Tomography (HRCT). Air trapping is defined as the percentage of lung voxels with mean attenuation below -856 Hounsfield units (HU).
Time Frame: Baseline, week 12.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent air trapping
Arm/Group | QBW251 300mg | Placebo
Number analyzed (Participants) | 19 | 18
percent air trapping
  Lung | -3.53 (7.534) | -0.95 (7.733)
  Lung, Left | -3.93 (7.176) | -0.89 (7.248)
  Lung, Left Lower Lobe | -4.27 (9.708) | -1.55 (7.486)
  Lung, Left Upper Lobe | -3.83 (7.220) | -0.78 (7.910)
  Lung, Right | -3.24 (8.280) | -0.98 (9.032)
  Lung, Right Lower Lobe | -3.57 (9.896) | -1.90 (11.666)
  Lung, Right Middle Lobe | -1.98 (10.362) | -0.80 (8.480)
  Lung, Right Upper Lobe | -2.09 (8.500) | 0.27 (8.934)
  Thirds, Left Lower | -5.40 (10.613) | -1.90 (8.111)
  Thirds, Left Middle | -3.56 (6.803) | -0.76 (6.659)
  Thirds, Left Upper | -2.84 (7.597) | -0.11 (9.272)
  Thirds, Right Lower | -4.52 (8.545) | -1.70 (10.890)
  Thirds, Right Middle | -3.28 (9.116) | -1.09 (8.218)
  Thirds, Right Upper | -1.84 (8.956) | 0.18 (10.107)

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until last dose of study treatment plus 7 days, up to a maximum duration of 99 days.
Groups:
- QBW251 300 mg b.i.d: QBW251 300 mg b.i.d
- Placebo: Placebo
- Total: Total
Arm/Group | QBW251 300 mg b.i.d | Placebo | Total
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/28 | 0/54
Serious Adverse Events (participants affected / at risk) | 2/26 | 0/28 | 2/54
Other Adverse Events (participants affected / at risk) | 12/26 | 5/28 | 17/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QBW251 300 mg b.i.d (N=26) | Placebo (N=28) | Total (N=54)
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QBW251 300 mg b.i.d (N=26) | Placebo (N=28) | Total (N=54)
Diarrhoea (Gastrointestinal disorders) | 4 | 0 | 4
COVID-19 (Infections and infestations) | 1 | 2 | 3
Nasopharyngitis (Infections and infestations) | 3 | 1 | 4
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 7
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-08-25): https://cdn.clinicaltrials.gov/large-docs/23/NCT04268823/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-23): https://cdn.clinicaltrials.gov/large-docs/23/NCT04268823/SAP_001.pdf